CLINICAL TRIAL: NCT06666231
Title: A Two-Center Randomized Controlled Trial
Brief Title: Comparison of Ultrasound-Guided Quadratus Lumborum Plane Block and External Oblique Intercostal Plane Block for Postoperative Analgesia After Laparoscopic Cholecystectomy: a Two-Center Randomized Controlled Trial
Acronym: A Two-Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Anesthesiology and Reanimation Spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTSsONER
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterior Quadratus Lumborum Plane Block (Active Comparator): After endotracheal intubation, patients in the supine position will be given a lateral tilt and the areas to be treated will be cleaned with surgical antiseptic solution. The convex USG probe will be covered in a sterile manner. Then, the sterile probe will be placed transversely on the crista iliaca. The probe will be directed cranially until the external oblique muscle, internal oblique muscle and transverse abdominis muscle are clearly visualized. The psoas major muscle and the transverse process of the vertebra will be visualized. The QL muscle will be visualized between the aponeuros of the transverse abdominis muscle and the psoas major muscle. A 20 G 100 mm block needle will be advanced from posterolateral to anteromedial using the "in-plane" technique. The needle will be directed between the QL muscle and the psoas major muscles. 20 ml of 0.25% bupivacaine (Buvasin®, Vem İlaç, Turkey) will be injected on each side between the fasciae of these two muscles and the LA distributio
  Interventions: Procedure: QL (quadratus lumborum) block administration
- External Oblique Intercostal Plane Block (Active Comparator): After endotracheal intubation, a 20-gauge 100 mm long block needle will be inserted at the T6-T7 level under USG guidance and bilateral EOIB will be applied with 20 cc of 0.25% Bupivacaine on each side under the external oblique intercostal muscle (total 40ml bilaterally).
  Interventions: Procedure: External Oblique Intercostal Plane Block

INTERVENTIONS:
Procedure: QL (quadratus lumborum) block administration — After endotracheal intubation, patients in the supine position will be given a lateral tilt and the areas to be treated will be cleaned with surgical antiseptic solution. The convex USG probe will be covered in a sterile manner. Then, the sterile probe will be placed transversely on the crista iliaca. The probe will be directed cranially until the external oblique muscle, internal oblique muscle and transverse abdominis muscle are clearly visualized. The psoas major muscle and the transverse process of the vertebra will be visualized. The QL muscle will be visualized between the aponeuros of the transverse abdominis muscle and the psoas major muscle. A 20 G 100 mm block needle will be advanced from posterolateral to anteromedial using the "in-plane" technique. The needle will be directed between the QL muscle and the psoas major muscles. 20 ml of 0.25% bupivacaine (Buvasin®, Vem İlaç, Turkey) will be injected on each side between the fasciae of these two muscles and the LA distribution
  Arms: Anterior Quadratus Lumborum Plane Block
Procedure: External Oblique Intercostal Plane Block — After endotracheal intubation, a 20-gauge 100 mm long block needle will be inserted at the T6-T7 level under USG guidance and bilateral EOIB will be applied with 20 cc of 0.25% Bupivacaine on each side under the external oblique intercostal muscle (total 40ml bilaterally).
  Arms: External Oblique Intercostal Plane Block

SUMMARY:
The primary aim of this study was to compare the postoperative analgesic efficacy of the Anterior Quadratus Lumborum Plane Block and the External Oblique Intercostal Plane Blocks used in laparoscopic cholecystectomy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo laparoscopic cholecystectomy and who meet the ASA I-II risk classification between the ages of 18-65 will be included.

Exclusion Criteria:

Patients who do not agree to participate in the study, who have an infection in the application area, who are allergic to local anesthesia, who have coagulopathy, who are morbidly obese (Body mass index (BMI)>35), who have a history of drug allergy, chronic pain, long-term opioid use and psychiatric illness, and who require emergency surgery are excluded from the study. will be left

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Postoperative 30.second,2 hours, 4 hours,12 hours,24 hours
  They will be numbered from 1 to 10. If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome

SECONDARY OUTCOMES:
Opioid use | postoperative 24 hours
  tramadol use
Riker Sedation Agitation Scale | Immediately after extubation
  7 Dangerous Agitation ... If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Patient satisfaction score | at the 24th postoperative hour
  Patients' satisfaction with the quality of pain management will be evaluated on the second postoperative day using the following scale: 1 = very unsatisfied; 2 = highly dissatisfied; 3 = medium; 4 = very satisfactory; 5 = very satisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Diyarbakır, kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No